CLINICAL TRIAL: NCT01386580
Title: An Open-label, Phase I/IIa, Dose Escalating Study of 2B3-101 in Patients With Solid Tumors and Brain Metastases or Recurrent Malignant Glioma.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BBB-Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2B3-101-CR-001
Record Dates: First submitted 2011-06-28; First posted 2011-07-01 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Brain Metastases; Lung Cancer; Breast Cancer; Melanoma; Malignant Glioma
Keywords: Brain Neoplasms; Neoplasm Metastasis; Neoplasms; Central Nervous System Neoplasms; Nervous System Neoplasms; Neoplasms by Site; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neoplastic Processes; Pathologic Processes
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Breast Neoplasms; Melanoma; Glioma; Neoplasm Metastasis; Neoplasms; Central Nervous System Neoplasms; Nervous System Neoplasms; Neoplasms by Site; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neoplastic Processes; Pathologic Processes | interventions — glutathione pegylated liposomal doxorubicin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2B3-101 Single Agent Dose Escalation (Experimental): Patients in single agent dose escalation arm will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. If tolerated, the infusion may then be completed over the next hour for a total infusion time of 90 minutes.
  Interventions: Drug: 2B3-101
- 2B3-101 in combination with trastuzumab (Experimental): HER2+ breast cancer patients with brain metastases will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. As long as 2B3-101 is well tolerated, the remaining 95% of the infusion could thereafter be administered over the next 60 min, resulting in a total infusion time of 90 minutes. The infusion of trastuzumab will then follow 30 minutes after the completion of the 2B3-101 infusion.
  Interventions: Drug: 2B3-101; Drug: Trastuzumab
- 2B3-101 solid tumor expansion (Experimental): Patients in the breast, Small Cell Lung Cancer and melanoma dose expansion arms will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. If tolerated, the infusion may then be completed over the next hour for a total infusion time of 90 minutes.
  Interventions: Drug: 2B3-101 50 mg/m2 every 3 weeks
- 2B3-101 glioma expansion (Experimental): Patients in the single agent glioma dose expansion arm will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. If tolerated, the infusion may then be completed over the next hour for a total infusion time of 90 minutes.
  Interventions: Drug: 2B3-101 60 mg/m2 every 4 weeks

INTERVENTIONS:
Drug: 2B3-101 — IV every 21 days
  Other Names: Glutathione pegylated liposomal doxorubicin hydrochloride
  Arms: 2B3-101 Single Agent Dose Escalation; 2B3-101 in combination with trastuzumab
Drug: Trastuzumab — IV every 21 days
  Other Names: Herceptin
  Arms: 2B3-101 in combination with trastuzumab
Drug: 2B3-101 60 mg/m2 every 4 weeks — IV every 28 days
  Other Names: Glutathione pegylated liposomal doxorubicin hydrochloride
  Arms: 2B3-101 glioma expansion
Drug: 2B3-101 50 mg/m2 every 3 weeks — IV every 21 days
  Other Names: Glutathione pegylated liposomal doxorubicin hydrochloride
  Arms: 2B3-101 solid tumor expansion

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics (PK) of 2B3-101 both as single agent and in combination with trastuzumab. Furthermore, the study will explore the preliminary antitumor activity of 2B3-101 as single agent in patients with with solid tumors and brain metastases or recurrent malignant glioma as well as in patients with various forms of breast cancer with and in combination with trastuzumab in HER2+ breast cancer patients with brain metastases.

DETAILED DESCRIPTION:
This is a Phase I/IIa, multicenter, open-label, dose-escalation study. The study will be conducted in 6 phases: "2B3-101 single agent dose-escalation phase", "a 2B3-101 with trastuzumab dose-escalation phase", "a Breast cancer brain metastases study-expansion phase","a Recurrent malignant glioma study-expansion phase", "a Melanoma brain metastases study- expansion phase" and "SCLC brain metastases study-expansion phase"

2B3-101 single agent dose-escalation phase.

In the 2B3-101 single Agent dose-escalation phase, female and male patients with solid tumors and brain metastases or recurrent malignant glioma will be enrolled. Patients will be assigned to a dose level cohort. - The starting dose will be 5 mg/m2, which is equal to 1/10 of the human equivalent dose of the LD10 of 2B3-101 in rats. A "3+3" dose-escalation design will be used. The study will investigate sequential cohorts consisting of 3-6 patients to be enrolled and treated at the applicable dose level. Planned dose levels for subsequent cohorts are 10, 20, 30, mg/m2 and steps of 10 mg/m2 thereafter. For more information on the dose escalation design and the increments, please see the dose escalation criteria section.

There will be no intra-patient dose escalation. Each treatment cycle consists of 21 days. Patients will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. If tolerated, the infusion may then be completed over the next hour for a total infusion time of 90 minutes. Blood samples will be taken on day 1, 2, 3, 5, 8 and 11 of cycle 1 and day 1, 8 and 15 of cycle 2 to assess the PK profile during the first 2 cycles. The dose limiting toxicity (DLT) observation period for each dose level will be cycle 1 (day 1 to day 21). Patients who do not complete the DLT observation period (cycle 1) for other reasons than a DLT will be replaced.

Once the MTD of 2B3-101 as single agent has been determined, the study will continue to the breast cancer brain metastases and recurrent malignant glioma dose expansion phases.

2B3-101 in combination with trastuzumab dose-escalation phase

In the 2B3-101 in combination with trastuzumab dose escalation phase, only patients with HER2+ breast cancer and brain metastases will be enrolled.

The patients will be assigned to a 2B3-101 dose level cohort. - The starting dose of 2B3-101 will be 40 mg/m2 every 3 weeks. This dose has been selected based upon safety information from patients treated with 2B3-101 at this dose level, as well as upon previous treatment with PEGylated liposomal doxorubicin in combinations trastuzumab (Chia et al 2006).

The dose-escalation will be conducted in steps of 10 mg/m2 up to the MTD level determined for 2B3-101 as single agent. The trastuzumab dose will remain fixed to a loading dose of 8 mg/kg at day 1 and 6 mg/kg every 3 weeks at the subsequent cycles throughout the determination of the MTD. Enrolment of HER2+ patients breast cancer patients in the "2B3-101 in combination with trastuzumab dose-escalation" phase of the study will be allowed in parallel with the determination of the MTD of 2B3-101 as single agent. A "3+3" dose-escalation design will be used. Thus, the study will investigate sequential cohorts of 3-6 patients, who will be enrolled and treated at the applicable dose levels.

No intra-patient dose-escalation will be allowed. Each treatment cycle consists of 21 days. All patients will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. As long as 2B3-101 is well tolerated, the remaining 95% of the infusion could thereafter be administered over the next 60 min, resulting in a total infusion time of 90 minutes. The infusion of trastuzumab will then follow 30 minutes after the completion of the 2B3-101 infusion. Blood samples will be taken on day 1, 2, 3, 5, 8 and 11 of cycle 1, on day 1, 8 and 15 of cycle 2 and if applicable on day 1 of cycle 3 and day 1 of cycle 4 to assess the PK profile of 2B3-101 during the first 4 cycles. The dose limiting toxicity (DLT) observation period will be cycle 1 (day 1 to day 21) at each individual dose level. Patients who do not complete the DLT observation period (cycle 1) for other reasons than a DLT will be replaced.

Breast cancer brain metastases expansion phase.

In the breast cancer brain metastases expansion phase, each treatment cycle consists of 21 days. Patients will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. If tolerated, the infusion may then be completed over the next hour for a total infusion time of 90 minutes. Blood samples will be taken on day 1, 2, 3, 5, 8 and 11 of cycle 1 on day 1, 8 and 15 of cycle 2 and if applicable on day 1 of cycle 3 and on day 1 of cycle 4 to assess the PK profile during the first 4 cycles.

Recurrent malignant glioma expansion phase.

In the recurrent malignant glioma expansion phase, each treatment cycle is 28 days long. Patients will receive a single IV dose of 2B3-101 on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose of 2B3-101 (in mg) should be infused slowly over the first 30 minutes. If tolerated, the infusion may then be completed over the next hour for a total infusion time of 90 minutes. Blood samples will be taken on day 1, 2, 3, 5, 8 and 11 of cycle 1, day 1, 8 and 15 of cycle 2 and if applicable on day 1 of cycle 3 and on day 1 of cycle 4 to assess the PK profile during the first 4 cycles.

SCLC brain metastases study arm of the expansion phase

In the SCLC brain metastases study arm of the expansion phase, each treatment cycle is 21 days long. Patients will receive a single IV dose of 2B3-101 at MTD determined for 2B3-101 as single agent on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose (in mg) should be infused slowly over the first 30 minutes. As long as 2B3-101 is well tolerated, the remaining 95% of the infusion could thereafter be administered over the next 60 minutes, resulting in a total infusion time of 90 minutes. Blood samples will be taken on day 1, 2, 3, 5, 8 and 11 of cycle 1, day 1, 8 and 15 of cycle 2 and if applicable on day 1 of cycle 3 and on day 1 of cycle 4 to assess the PK profile during the first 4 cycles.

Melanoma brain metastases study arm of the expansion phase

In the melanoma brain metastases study arm of the expansion phase, each treatment cycle is 21 days long. Patients will receive a single IV dose of 2B3-101 at MTD determined for 2B3-101 as single agent in the dose escalation phase on day 1 of each cycle. In order to minimize the risk of infusion reactions 5% of the total dose (in mg) should be infused slowly over the first 30 minutes. As long as 2B3-101 is well tolerated, the remaining 95% of the infusion could thereafter be administered over the next 60 minutes, resulting in a total infusion time of 90 minutes. Blood samples will be taken on day 1, 2, 3, 5, 8 and 11 of cycle 1, day 1, 8 and 15 of cycle 2 and if applicable on day 1 of cycle 3 and on day 1 of cycle 4 to assess the PK profile during the first 4 cycles.

For all stages a patient will stay on treatment until disease progression, unacceptable toxicity, or discontinuation for any other reason.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Measurable intracranial disease by MRI.
3. ECOG Performance Status ≤ 2.
4. Estimated life expectancy of at least 8 weeks.
5. Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ grade 2 (as defined by CTCAE version 4.0).
6. No evidence of (cortical) cognitive impairment as defined by a Mini-Mental Status Exam (MMSE) score ≥ 25/30.
7. Written informed consent according to local guidelines.

In addition to the above listed eligibility criteria, the following criteria are applicable:

8.

* 2B3-101 single agent dose-escalation phase:

  1. Patients with pathologically confirmed diagnosis of advanced, recurrent solid tumors and unequivocal evidence of brain metastases that are refractory to standard therapy or for whom no standard therapy exists or with unequivocal evidence of newly diagnosed untreated brain metastases and controlled extracranial disease which per the multi-disciplinary team decision do not require immediate radiotherapy, surgery or standard systematic chemotherapy. Brain metastases may be stable, progressive, symptomatic or asymptomatic brain metastasis/es. Stable or decreasing dosage of steroids (e.g. dexamethasone) for 7 days prior to baseline MRI or non-enzyme inducing anti-epileptic drugs is allowed.

     Or -
  2. Patients with pathology confirmed diagnosis of advanced, recurrent primary malignant (grade III and IV) glioma that are refractory to standard therapy or for whom no standard therapy exists. Stable or decreasing dosage of steroids (e.g. dexamethasone) for 7 days prior to baseline MRI or non-enzyme inducing anti-epileptic drugs are allowed.
* 2B3-101 in combination with trastuzumab dose escalation phase:

Patients with histologically-confirmed HER2-positive (IHC 3+ or fluorescence in situ hybridization [FISH] amplified; by clinical assay on either primary or metastatic tumor) adenocarcinoma of the breast with unequivocal evidence of brain metastases that are refractory to standard therapy or for which no standard therapy exist or with unequivocal evidence of newly diagnosed untreated brain metastases and controlled extracranial disease which per the multi-disciplinary team decision do not require immediate radiotherapy, surgery or standard systematic chemotherapy can be included to this escalation phase as well.

- Breast cancer brain metastases expansion phase:

1. Patients with pathologically confirmed diagnosis of advanced, recurrent breast cancer with at least one progressive and/or new metastatic brain lesion, that are refractory to standard therapy or for whom no standard therapy exist. Brain metastases may be stable, progressive, symptomatic or asymptomatic brain metastasis/es. Stable or decreasing dosage of steroids (e.g. dexamethasone) for 7 days prior to baseline MRI or non-enzyme inducing anti-epileptic drugs is allowed.

   Or -
2. Patients with pathologically confirmed diagnosis of advanced breast cancer with newly diagnosed, untreated, brain metastases and controlled extracranial disease which per the multi-disciplinary team decision do not require immediate radiotherapy, surgery or standard systematic chemotherapy.

SCLC brain metastases study arm of the expansion phase:

1. Patients with pathologically confirmed diagnosis of advanced, recurrent SCLC with at least one progressive and/or new metastatic brain lesion that are refractory to standard therapy or for whom no standard therapy exist. Stable or decreasing dosages of steroids (e.g. dexamethasone) for 7 days prior to baseline MRI and/or use of non-enzyme inducing anti-epileptic drugs are allowed.

   Or
2. Patients with pathologically confirmed diagnosis of advanced SCLC with newly diagnosed, untreated, brain metastases and controlled extracranial disease which per the multi-disciplinary team decision do not require immediate radiotherapy, surgery or standard systematic chemotherapy.

Melanoma brain metastases study arm of the expansion phase:

1. Patients with pathologically confirmed diagnosis of advanced, recurrent melanoma with at least one progressive and/or new metastatic brain lesion that are refractory to standard therapy or for whom no standard therapy exist. Stable or decreasing dosages of steroids (e.g. dexamethasone) for 7 days prior to baseline MRI and/or use of non-enzyme inducing anti-epileptic drugs are allowed.

   Or
2. Patients with pathologically confirmed diagnosis of advanced melanoma with newly diagnosed, untreated, brain metastases and controlled extracranial disease which per the multi-disciplinary team decision do not require immediate radiotherapy, surgery or standard systematic chemotherapy.

Recurrent malignant glioma study arm of the expansion phase:

1. 7 patients with histologically proven glioma grade IV, which is progressive following first line treatment with surgery or biopsy followed by fractionated radiotherapy with concurrent temozolomide-containing chemotherapy.

   and
2. 7 patients with recurrent histologically confirmed malignant (WHO grade III and IV) glioma or histologically confirmed low-grade (WHO grade II) glioma with radiographic evidence of malignant transformation by MRI, that are refractory to standard therapy, or for whom no standard therapy exists or do not require immediate standard therapy per the multi-disciplinary team decision. Patients in both groups should have stable or decreasing dosage of steroids (e.g. dexamethasone) for a minimum of 7 days prior to baseline MRI. Non-enzyme inducing anti-epileptic drugs are allowed

   Exclusion Criteria.
   * Prior Treatment. 1. Less than 1 week since the last treatment of lapatinib, less than 2 weeks since the last treatment of vemurafenib, less than 4 weeks since the last treatment of chemotherapy, biological therapy, immunotherapy and systemic radiotherapy (except palliative radiation delivered to <20% of bone marrow), less than 8 weeks for cranial radiotherapy, and less than 6 weeks for nitrosoureas and mitomycin C.

     2. Patients that have received a maximum cumulative dose of free (i.e., non-liposomal) or liposomal doxorubicin > 360mg/m2 or free epirubicin > 600mg/m2.
   * Current Treatment. 3. Current or recent (within 30 days of first study treatment) treatment with another investigational drug or participation in another investigational study.
   * Hematology, coagulation and biochemistry. 4. Inadequate bone marrow function: Absolute Neutrophil Count (ANC): < 1.5 x 109/L, or platelet count < 100 x 109/L or hemoglobin < 6 mmol/L.

     5. Inadequate liver function, defined as:

     • Serum (total) bilirubin > 1.5 x the ULN for the institution if no liver metastases (> 2 x ULN in patients with liver metastases);

     • ASAT or ALAT > 2.5 x ULN if no liver metastases (> 4 x ULN in patients with liver metastases);
     * Alkaline phosphatase levels > 2.5 x ULN if no liver metastases (> 5 x ULN in patients with liver metastases, or > 10 x ULN in patients with bone metastases).

       6. Inadequate renal function, defined as:
     * Serum creatinine > 1.5 x ULN.
   * Other. 7. Leptomeningeal carcinomatosis as the only site of CNS involvement. 8. Pregnancy or lactation. Serum pregnancy test to be performed within 7 days prior to study treatment start, or within 14 days followed by a confirmatory urine pregnancy test within 7 days prior to study treatment start.

     9. For female subjects of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male subjects who are not surgically sterile or with female partners of childbearing potential: absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel).

     10. Major surgical procedure (including open biopsy, excluding central line IV and portacath) within 28 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment.

     11. Grade 3 or 4 motor, sensory, or cranial neuropathy symptoms (as defined by CTCAE version 4.0).

     12. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100mm Hg).

     13. Clinically significant (i.e. active) cardiovascular disease defined as:

     • Stroke within ≤ 6 months prior to day 1;

     • Transient Ischemic Attack (TIA) within ≤ 6 months prior to day 1;

     • Myocardial infarction within ≤ 6 months prior to day 1;

     • Unstable angina;
     * New York Heart Association (NYHA) Grade II or greater Congestive Heart Failure (CHF);
     * Serious cardiac arrhythmia requiring medication;
     * Clinically relevant pathologic findings in ECG. 14. Left Ventricle Ejection Fraction (LVEF) by MUGA or ECHO < 55% for patients receiving 2B3-101 in combination with trastuzumab. For patients receiving single agent 2B3-101 treatment. Left Ventricle Ejection Fraction (LVEF) by MUGA or ECHO < 50%.

       15. Known hypersensitivity to any of the study drugs excipients (e.g. doxorubicin, PEG or GSH).

       16. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, physical examination or laboratory findings) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of intravenously administered 2B3-101 in patients with advanced solid tumors and metastatic brain cancer or recurrent malignant glioma. | 16 months
To identify the maximum tolerated dose (MTD) of of intravenously administered 2B3-101 in patients with advanced solid tumors and metastatic brain cancer or recurrent malignant glioma. | 16 months
To assess the safety and tolerability of intravenously (IV) administered 2B3-101 in combination with trastuzumab, in patients with HER2+ breast cancer with brain metastases | 9 months
To identify the maximum tolerated dose (MTD) of of intravenously administered 2B3-101 in combination with trastuzumab in patients with HER2+ breast cancer with brain metastases | 9 months

SECONDARY OUTCOMES:
Examine the pharmacokinetics (PK) in plasma of intravenously administered 2B3-101 in terms of Cmax, Vss, T1/2, AUC, CL; | 16 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on brain metastases secondary to breast cancer in terms of objective response rate. | 16 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on brain metastases secondary to breast cancer in terms of duration of response. | 16 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on recurrent malignant glioma in terms of objective response rate. | 16 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on recurrent malignant glioma in terms of duration of response. | 16 months
Examine the pharmacokinetics (PK) in plasma of intravenously administered 2B3-101 in combination with trastuzumab in terms of Cmax, Vss, T1/2, AUC, CL; | 9 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 in combination with trastuzumab on brain metastases secondary to HER2+ breast cancer in terms of objective response rate. | 9 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 in combination with trastuzumab on brain metastases secondary to HER2+ breast cancer in terms of duration of response. | 9 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on brain metastases secondary to SCLC cancer in terms of objective response rate. | 6 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on brain metastases secondary to melanoma in terms of objective response rate. | 6 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on brain metastases secondary to SCLC cancer in terms of duration of response. | 6 months
Obtain preliminary information on the clinical anti-tumor activity of intravenously administered 2B3-101 on brain metastases secondary to melanoma in terms of duration of response. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: J. Veeneman, PhD, Study Director — BBB Therapeutics
Locations (10):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Jules Bordet Institute, Brussels
- France (2):
  - Institut Curie, Paris, Paris Cedex 05
  - Institut Gustave Roussy, Villejuif, Val de Marne
- Netherlands (5):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Vrije Universiteit medisch centrum (Vumc), Amsterdam
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus MC, Rotterdam